CLINICAL TRIAL: NCT03416699
Title: Chinese Transanal Total Mesorectal Excision Registry Collaborative: A Nationwide Registry Study
Brief Title: Chinese TaTME Registry Collaborative
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Ruijin Hospital (Other); Peking Union Medical College Hospital (Other); Peking University Cancer Hospital & Institute (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shengjing Hospital (Other); Huashan Hospital (Other); Guangdong Dongguan Kanghua Hospital (Unknown); Guangdong Provincial People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Nanchong Central Hospital (Other Government); Sino-Japanese Friendship Hospital of Jilin University (Unknown); Koo Foundation Sun Yat-Sen Cancer Center (Other); Shangdong Linzi District People's Hospital (Unknown); Peking University People's Hospital (Other); Nantong University (Other); Liaoning Cancer Hospital & Institute (Other); The First Hospital of Jilin University (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Nanjing PLA General Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Sichuang Zigong First People's Hospital (Unknown); Beijing Chao Yang Hospital (Other); Peking University Third Hospital (Other); Jinhua Central Hospital (Other); Beijing Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Tianjin Medical University General Hospital (Other); LanZhou University (Other); Chinese PLA General Hospital (Other); Cancer Hospital of Guizhou Province (Other); First Hospital of China Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, assistant dean, professor, Beijing Friendship Hospital
Other Study IDs: CTRC
Record Dates: First submitted 2018-01-01; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Rectal Cancer
Keywords: Transnal Total Mesorectal Excision; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total mesorectal excision (TME) is the gold standard procedure for treating rectal cancer. However, in patients with obesity, prostate hypertrophy, low located tumor or/and pelvic stenosis, the traditional laparoscopic or open surgery is not easy to conduct. Transanal total mesorectal excision (TaTME) might serve as a better procedure for these patients, for it might ease the dissection of the low mesorectum. So far, several studies have showed the promising results of TaTME, but the multi-center data in China is still lacking. This nationwide registry study included more than 30 Chinese hospitals, aiming at obtaining data on the safety and efficacy of this procedure in Chinese patients with rectal cancer and encouraging future research in this field.

ELIGIBILITY:
Inclusion Criteria:

* malignant or benign neoplasms of the rectum
* the lower edge of the tumor from the anal margin less than 10cm according to MRI or rigid endoscopy
* tolerable to surgery
* be able to understand and willing to participate in this registry with signature

Exclusion Criteria:

* patients requiring emergency surgery such as obstruction，perforation and bleeding
* tumor involving adjacent organs, anal sphincter, or levator ani muscle
* muti-focal colorectal cancer
* preoperative poor anal function, anal stenosis, anal injury, or fecal incontinence
* history of inflammatory bowel disease or familial adenomatous polyposis
* can not tolerate the surgery
* history of serious mental illness
* pregnancy or lactating women
* preoperative uncontrolled infection
* the researchers believe the patients should not enrolled in

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with middle-lower rectal neoplasms who are suitable and willing to accept TaTME procedure and also agree with the registry
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Positive rate of circumferential resection margin (CRM) of the specimens | 10 days after surgery
  Circumferential resection margin (CRM) is the distance between the deepest point of tumor in the primary cancer and the margin of resection in the retroperitoneum or mesentery by pathological examination. CRM 0-1mm is defined as positive, while >1mm is negative.
The grade score of the specimens integrity | 10 days after surgery
  shows the quality of the specimens: grade 1 is bad gross specimen which means incomplete mesorectum and pelvic fascia, and muscle layer can be see >5mm; grade 3 is high quality gross specimen, which means the specimen is cylindrical, mesorectum and pelvic fascia are complete; grade 2 is between 1and 3.

SECONDARY OUTCOMES:
local recurrence rate | 3 years after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
disease free survival rate | 3-year after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
overall survival rate | 3-year after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
the incidence of postoperative complications | 30 days after surgery
  the incidence of postoperative complications after transanal total mesorectal excision.
the severity of postoperative complication assessed by Clavien Dindo grade | 30 days after surgery
  the severity of postoperative complication after transanal total mesorectal assessed by Clavien Dindo grade
the grade of anastomotic leakage | 30 days after surgery
  the grade of anastomotic leakage for patients who develop anastomotic leakage after transanal total mesorectal excision assessed by the grading system proposed by International Study Group of Rectal Cancer (ISREC).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

REFERENCES:
- [Derived] Li Q, Yang X, Teng Q, Guo Q, Qin L, Lv Z, Zhou D, Ren M. Reasonable Collocation of Two Different Functional 3D Laparoscopes May Improve the Efficiency of Transanal Total Mesorectal Excision Surgery Using a Synchronous Two-Team Approach? J Laparoendosc Adv Surg Tech A. 2023 Feb;33(2):194-199. doi: 10.1089/lap.2022.0326. Epub 2022 Jul 22. PMID 35867023